CLINICAL TRIAL: NCT07248579
Title: Cross-Cultural Adaptation and Psychometric Validation of the Turkish Version of the Pregnancy-Specific Anxiety Tool (PSAT-TR) Among Pregnant Women
Brief Title: Turkish Validation of the Pregnancy-Specific Anxiety Tool (PSAT)
Acronym: PSAT-TR
Status: Completed | Type: Observational
Sponsor: Havva Betül Bacak (Other Government)
Collaborators: İstanbul Gaziosmanpaşa Training and Research Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Havva Betül Bacak, M.D, Gaziosmanpasa Research and Education Hospital
Organization: Gaziosmanpasa Research and Education Hospital (Other Government)
Other Study IDs: psat turkish validation
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy-related Anxiety; Antenatal Anxiety; Perinatal Mental Health
Keywords: Pregnancy-Specific Anxiety Tool (PSAT); PSAT-TR; Pregnancy anxiety; Antenatal anxiety; Perinatal mental health; Scale validation; Psychometric analysis; Reliability and validity; Turkish adaptation; Cross-sectional study

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant Women: Pregnant women aged 18 years and older who attended routine antenatal care at Gaziosmanpasa Training and Research Hospital between September and October 2025. Participants completed three self-report questionnaires: the Turkish version of the Pregnancy-Specific Anxiety Tool (PSAT-TR), the State-Trait Anxiety Inventory-State (STAI-State), and the Pregnancy-Related Anxiety Questionnaire-Revised 2 (PRAQ-R2). No medical, pharmacological, or procedural intervention was applied.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Administration of three self-report questionnaires for psychometric validation: the Turkish version of the Pregnancy-Specific Anxiety Tool (PSAT-TR), the State-Trait Anxiety Inventory-State (STAI-State), and the Pregnancy-Related Anxiety Questionnaire-Revised 2 (PRAQ-R2). Participants completed the questionnaires during a single antenatal clinic visit. No medical, pharmacological, or procedural intervention was applied.
  Other Names: PSAT-TR; STAI-State; PRAQ-R2

SUMMARY:
The Pregnancy-Specific Anxiety Tool (PSAT) is a newly developed instrument designed to assess anxiety specific to pregnancy across multiple domains. This methodological, cross-sectional study aims to adapt the PSAT into Turkish and to evaluate its psychometric properties among pregnant women in Turkey. The study evaluates the reliability and validity of the Turkish version (PSAT-TR) through internal consistency, factor analysis, and criterion validity analyses using the State-Trait Anxiety Inventory-State (STAI-State) and the Pregnancy-Related Anxiety Questionnaire-Revised 2 (PRAQ-R2). Data were collected from pregnant women attending antenatal care at Gaziosmanpasa Training and Research Hospital. The study hypothesizes that the Turkish version of PSAT is a valid and reliable instrument to assess pregnancy-related anxiety in the Turkish population.

DETAILED DESCRIPTION:
This methodological, cross-sectional, single-center study was conducted to adapt the Pregnancy-Specific Anxiety Tool (PSAT) into Turkish and to evaluate its psychometric properties. The PSAT is a 33-item scale developed by Harrison et al. (2023) to assess pregnancy-specific anxiety across six domains: (1) severity of anxiety, (2) health and well-being of the baby, (3) labor and maternal well-being, (4) postpartum concerns, (5) career and financial issues, and (6) social support.

The adaptation process followed internationally accepted guidelines, including forward and backward translation, expert committee review, and pilot testing to ensure linguistic and cultural equivalence. The final Turkish version (PSAT-TR) was administered to pregnant women aged 18 years and older, between 12 and 40 weeks of gestation, who attended routine antenatal follow-up at Gaziosmanpasa Training and Research Hospital. Participants provided written informed consent, and the study was approved by the hospital's Non-Interventional Clinical Research Ethics Committee (Approval No: 2025/-, Date: September 17, 2025).

Data were collected between September and October 2025. A total of approximately 300 participants completed the PSAT-TR, STAI-State, and PRAQ-R2 questionnaires. Internal consistency reliability was assessed using Cronbach's alpha coefficients. Construct validity was evaluated through exploratory and confirmatory factor analyses. Criterion validity was examined via correlations between PSAT-TR, STAI-State, and PRAQ-R2 scores. Receiver Operating Characteristic (ROC) analysis was used to determine optimal PSAT cut-off values based on STAI-State (≥40) and PRAQ-R2 (≥30) reference points.

The study aims to provide a culturally adapted, valid, and reliable tool to measure pregnancy-specific anxiety in Turkish-speaking populations. This tool may facilitate early identification of anxiety symptoms and inform preventive strategies in perinatal mental health care.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18-45 years
* Currently in 12-40 weeks of gestation
* Able to read and understand Turkish
* Voluntarily agreed to participate and provided written informed consent
* Attending routine antenatal care at Gaziosmanpasa Training and Research Hospital

Exclusion Criteria:

* Presence of a diagnosed psychiatric disorder
* Current use of psychiatric medication
* High-risk pregnancy or severe obstetric complication
* Inability to complete self-report questionnaires due to cognitive or literacy limitations

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consisted of pregnant women aged 18-45 years who attended routine antenatal follow-up at Gaziosmanpasa Training and Research Hospital. Participants were healthy, low-risk pregnancies without any known psychiatric or obstetric complications.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2025-09-17 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
Psychometric validity and reliability of the Turkish version of the Pregnancy-Specific Anxiety Tool (PSAT-TR) | Within 1 month after data collection
  The primary outcome is to assess the psychometric properties of the Turkish version of the Pregnancy-Specific Anxiety Tool (PSAT-TR) through exploratory and confirmatory factor analysis, internal consistency (Cronbach's alpha), and test-retest reliability. Validity is examined by comparing PSAT-TR scores with the State-Trait Anxiety Inventory-State (STAI-State) and the Pregnancy-Related Anxiety Questionnaire-Revised 2 (PRAQ-R2).

SECONDARY OUTCOMES:
Determination of optimal PSAT-TR cut-off values for pregnancy-related anxiety | Within 1 month after primary data analysis
  The secondary outcome is to determine optimal cut-off scores of the PSAT-TR for detecting elevated pregnancy-related anxiety. Receiver Operating Characteristic (ROC) analysis will be performed using STAI-State (≥40) and PRAQ-R2 (≥30) as external reference standards to evaluate sensitivity, specificity, and area under the curve (AUC) values.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Gaziosmanpaşa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participant-level data are not intended for public sharing due to ethical and institutional restrictions.

REFERENCES:
- [Result] Bayrampour H, Hohn RE, Tamana SK, Sawatzky R, Janssen PA, Bone JN, Fairbrother N, Joseph KS. Pregnancy-Specific Anxiety Tool (PSAT): Instrument Development and Psychometric Evaluation. J Clin Psychiatry. 2023 Apr 19;84(3):22m14696. doi: 10.4088/JCP.22m14696. PMID 37074299